CLINICAL TRIAL: NCT02588365
Title: Randomized Controlled Trial of Executive Function Training in Children With or At-risk for Attention-Deficit/Hyperactivity Disorder (ADHD) and Executive Function (EF) Impairment
Brief Title: Brain Training in Children With/At-risk for Attention-Deficit/Hyperactivity Disorder and Executive Function Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Irene M. Loe, MD, Principal Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 30874-2
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; executive function; preschool
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Training; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Brain Training (Active) (Experimental): The children in this arm receive one type of "Brain Training" with online computer games that actively matches their skill level.
  Interventions: Behavioral: Brain Training (Active)
- Brain Training (Passive) (Experimental): The children in this arm receive one type of "Brain Training" with online computer games that are at a consistent level.
  Interventions: Behavioral: Brain Training (Passive)
- Cross-over (Experimental): Following completion of the 6-month follow-up sessions after completion of "Brain Training", each group is allowed to cross-over to the other arm of "Brain Training" (open-label extension).
  Interventions: Behavioral: Brain Training (Active or Passive)

INTERVENTIONS:
Behavioral: Brain Training (Active) — Online computer games targeting attention, EF, and problem-solving
  Arms: Brain Training (Active)
Behavioral: Brain Training (Passive) — Online computer games targeting attention, EF, and problem solving
  Arms: Brain Training (Passive)
Behavioral: Brain Training (Active or Passive) — Online computer games targeting attention, EF, and problem solving
  Arms: Cross-over

SUMMARY:
The purpose of this study is to determine if different forms of child-friendly, computer-based puzzles and games ("brain training") targeting executive function (EF) skills (i.e., thinking, problem-solving) result in improvements in EF in preschool children with or at-risk for Attention-Deficit/Hyperactivity Disorder (ADHD) and EF problems. The investigators hypothesize that children receiving active "brain training" will show greater improvements in EF and related skills immediately after treatment than children receiving passive "brain training." The investigators are also interested in whether any improvements in EF and related skills occur or are maintained at 3 and 6 months after completion of brain training.

DETAILED DESCRIPTION:
* Investigators will talk to you by telephone to determine if your child might be eligible for the study.
* Children complete two baseline testing sessions to evaluate executive function (EF) and related skills
* Parents complete a packet of information, including questionnaires about the child's behavior, EF, and functional skills.
* After completion of the baseline testing, we will inform you of eligibility for the "Brain Training" phase.
* During "Brain Training" children play online computer games for 25-30 minutes/day (can range from 15-45 minutes/day depending on your child's attention, training version received, number and length of breaks needed), 5 days a week, for 5-7 weeks to complete a total of 25 sessions.
* Children return for 3 more time points, immediately after the completion of "Brain Training" (1 session), and also at 3 months (1 session) and 6 months (2 sessions) after completion of "Brain Training."

ELIGIBILITY:
Inclusion Criteria:

* Age 4 or 5 years
* Born Full term (37 weeks gestation or greater)
* Diagnosis of ADHD or high ADHD symptoms (T-score 60 or greater on standardized behavior questionnaire)
* Able to comprehend task instructions

Exclusion Criteria:

* Major neurosensory impairment (ie blind, deaf) that interferes with testing
* Genetic syndrome
* Inability to comprehend task instructions

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Change fro baseline on Executive Function Composite Measure at 2 months | 2 months
  EF composite measured post "Brain Training"

SECONDARY OUTCOMES:
Change from baseline on Executive Function Composite measure at 5 months | 5 months
  EF composite measured 3-months post "Brain Training" and 5 months from baseline
Change from baseline on Executive Function Composite measure at 8 months | 8 months
  EF composite measured 6-months post "Brain Training" and 8 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Irene M Loe, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States